CLINICAL TRIAL: NCT00858117
Title: A Phase II Trial of Alemtuzumab (Campath-1H) and Rituximab (Rituxan) in Patients With Previously Untreated CLL
Brief Title: A Phase II Trial of Alemtuzumab and Rituximab in Patients With Previously Untreated CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04H6; NU 04H6 (Other: Northwestern University); STU00004494 (Other: Northwestern University IRB)
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab and Rituximab (Experimental): Administration of Alemtuzumab combined with Rituximab to test the feasibility of combining these two monoclonal antibodies as a first line therapy in patients with B-cell chronic lymphocytic leukemia.
  Interventions: Biological: Alemtuzumab; Biological: Rituximab

INTERVENTIONS:
Biological: Alemtuzumab — Alemtuzumab administered subcutaneously 30mg per day, 3 days per week for 18 weeks
  Other Names: Campath-1H
Biological: Rituximab — Rituximab administered intravenously at 375mg/m2 every 2 weeks for 18 weeks
  Other Names: Rituxan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab and rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving alemtuzumab together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of giving alemtuzumab together with rituximab and to see how well it works in treating patients with previously untreated B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the response rate in patients with previously untreated B-cell chronic lymphocytic leukemia treated with alemtuzumab and rituximab.
* To evaluate the toxicity of alemtuzumab and rituximab in these patients.

OUTLINE: Patients receive alemtuzumab subcutaneously on days 1, 3, and 5 in weeks 1-18 and rituximab IV on day 1 in weeks 3, 5, 7, 9, 11, 13, 15, and 17 in the absence of disease progression or unacceptable toxicity.

Peripheral blood and bone marrow samples are collected periodically for laboratory biomarker studies. Samples are analyzed for surface markers (e.g., CD3, CD4, CD8, CD10, CD19, CD20, CD25, CD38, CD52, Zap-70) and IgVH by PCR, flow cytometry, and FISH. Samples are also analyzed for alemtuzumab and anti-alemtuzumab antibody levels by flow cytometry.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL)*, as defined by the following criteria:

  * Peripheral blood absolute lymphocyte count > 5,000/mm³
  * Small- to moderate-size lymphocytes with < 55% prolymphocytes, atypical lymphocytes, or lymphoblasts
  * Phenotypically characterized B-CLL expressing CD20 and CD52, as defined by the following:

    * Predominant population of cells share B-cell antigens with CD-5 in the absence of other pan-T-cell markers (e.g., CD-3, CD-2)
    * B-cell expresses either lambda or kappa light chains
    * Surface immunoglobulin with low-cell surface density expression NOTE: *Presence of splenomegaly, hepatomegaly, or lymphadenopathy are not required for the diagnosis of CLL
* Requires therapy, as indicated by ≥ 1 of the following criteria:

  * Unintentional weight loss > 10% within the past 6 months
  * Extreme fatigue (i.e., ECOG performance status 2)
  * Fevers > 100.5°F for 2 weeks without evidence of infection
  * Night sweats without evidence of infection
  * Evidence of progressive marrow failure as manifested by the development of or worsening of anemia (hemoglobin < 10 g/dL) and/or thrombocytopenia (platelet count < 100,000/mm³)
  * Massive (i.e., > 6 cm below left costal margin) or progressive splenomegaly
  * Massive nodes/clusters (> 5 cm), progressive symptomatic adenopathy, or adenopathy resulting in end-organ damage
  * Progressive lymphocytosis with an increase of > 50% over 2 months or an anticipated doubling time < 6 months
* Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease is not sufficient for eligibility

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,000/mm³*
* Platelet count ≥ 50,000/mm³*
* Hemoglobin ≥ 10 g/dL*
* Serum creatinine ≤ 2.0 mg/dL OR creatinine clearance > 40 mL/min
* Bilirubin < 2 mg/dL
* AST and ALT ≤ 2 times normal (unless secondary to tumor infiltration/lymphadenopathy)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No active autoimmune anemia or thrombocytopenia
* No active infection requiring oral or intravenous antibiotics
* No second malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix, unless curatively treated ≥ 2 years ago NOTE: *If cytopenias are due to degree of bone marrow involvement, patient may be eligible at the discretion of the principal investigator.

PRIOR CONCURRENT THERAPY:

* Prior corticosteroid therapy allowed
* No prior cytotoxic therapy (other than corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09-26 (Actual); Primary Completion 2010-03-17 (Actual); Study Completion 2013-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Frankfurt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on 29th March 2005 with the first patient starting treatment 26th September 2005 and an accrual goal of 30 patients. The study closed to further enrollment on the 26th October 2009 with 30 patients treated on study.
Groups:
- Alemtuzumab and Rituximab: Administration of Alemtuzumab combined with Rituximab to test the feasibility of combining these two monoclonal antibodies as a first line therapy in patients with B-cell chronic lymphocytic leukemia.
  Alemtuzumab: Alemtuzumab administered subcutaneously 30mg per day, 3 days per week for 18 weeks
  Rituximab: Rituximab administered intravenously at 375mg/m2 every 2 weeks (starting week 3) for 18 weeks
Period: Treatment on Study
Arm/Group | Alemtuzumab and Rituximab
Started | 30
Completed 18 Weeks of Treatment | 28
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 2
Period: Follow up for 5 Years
Arm/Group | Alemtuzumab and Rituximab
Started | 30 (All patients who receive at least one dose of drug under the protocol go into follow up for survival)
Completed | 17
Not Completed | 13
Not completed — Death | 4
Not completed — No further data collected for study | 9

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab and Rituximab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Treated With Alemtuzumab and Rituximab Combination With a Response (CR or PR) Assessed by NCI-WG 1996 Criteria With Lymph-adenopathy and Organomegaly Measured During Physical Examination
Description: Response rate (complete remission(CR) + partial remission(PR)) will be, assessed by NCI-WG 1996 criteria with lymphadenopathy and organomegaly measured during physical examination.
  CR=Absence of lymphadenopathy and constitutional symptoms, Normal CBC (leukocytes ≥ 1500/μl, Platelets >100,000/μl, Hemoglobin > 11.0 gm/dl), peripheral blood lymphocytes ≤ 4,000/μl.The marrow sample must be at least normocellular with < 30% of nucleated cells being lymphocytes.
  PR=absence of constitutional symptoms, ≥ 50% decrease in peripheral blood lymphocyte count from the pretreatment baseline value, ≥ 50% reduction in lymphadenopathy, ≥ 50% reduction in size of liver and/or spleen and one of the following:
  polymorphonuclear leukocytes ≥ 1,500/μl or 50% improvement over baseline platelets > 100,000/μl or 50% improvement over baseline or hemoglobin > 11.0 gm/dl or 50% improvement over baseline without transfusions
Time Frame: At week 9, and post-18 weeks then every 3 months for a year and up every 6 months for up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab and Rituximab
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: Number of Patients Treated With Alemtuzumab and Rituximab Combination With Response (CR or PR) Assessed by NCI-WG 1996 Criteria With Measurements of the Lymph Nodes and Spleen Size by CT Scans
Description: Response rate (complete remission(CR) + partial response(PR)) will be assessed by NCI-WG 1996 criteria with measurements of the lymph nodes and spleen size by CT scans. Best response at any timepoint is captured below.
  CR= absence of significant lymphadenopathy (e.g. lymph nodes > 1.5 cm in their greatest transverse diameter) and no hepatomegaly or splenomegaly.
  PR=reduction in lymphadenopathy as defined by the following: (a) a decrease in lymph node size by 50% or more either in the sum products of up to six lymph nodes, or in the largest diameter of the enlarged lymph node(s) detected prior to therapy; (b) no increase in any lymph node, and no new enlarged lymph node; in small lymph nodes (< 2cm), an increase of less than 25% was not considered to be significant and a reduction in the noted pretreatment enlargement of the spleen or liver by 50% or more.
Time Frame: At week 9, and post-18 weeks then every 3 months for a year and up every 6 months for up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab and Rituximab
Number analyzed (Participants) | 30
Participants | 21

3. Secondary Outcome: Toxicity of the Study Medications, Alemtuzumab and Rituximab
Description: Toxicity data will be collected at visits during 18 weeks of treatment and include adverse events considered at least possibly related to either study drugs (Alemtuzumab and Rituximab) and graded 3-5 using CTCAE 3.0.
  In general grading is as follows:
  Grade 1=mild Grade 2=moderate Grade 3=severe Grade 4=life threatening Grade 5=death Reported below are the number of patients who experienced each event
Time Frame: During treatment, 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab and Rituximab
Number analyzed (Participants) | 30
Participants
  Neutropenia | 9
  Thrombocytopenia | 2
  Infection | 2
  Renal toxicity | 1
  Skin rash | 1
  Fatigue | 1

4. Post Hoc Outcome: Best Response in Patients Treated With Alemtuzumab and Rituximab Combination Assessed by NCI-WG 1996 Criteria With Lymphadenopathy and Organomegaly Measured During Physical Examination
Description: Patients best response to treatment as defined in general as:
  Complete Remission=Absence of lymphadenopathy and constitutional symptoms, Normal CBC, peripheral blood lymphocytes ≤ 4,000/μl.The marrow sample must be at least normocellular with < 30% of nucleated cells being lymphocytes.
  Partial Remission=absence of constitutional symptoms, ≥50%decrease in peripheral blood lymphocyte count, ≥50%reduction in lymphadenopathy, ≥50%reduction in liver and/or spleen size & 1 of the following:
  polymorphonuclear leukocytes ≥ 1,500/μl or 50% improvement over baseline, platelets >100,000/μl or 50%improvement over baseline, hemoglobin > 11.0 gm/dl or 50% improvement over baseline without transfusions. Stable Disease=Do not meet criteria for complete/partial remission or progressive disease.
  Progressive Disease= ≥50%increase ≥2 lymph nodes or ≥50% increase in absolute no. of circulating lymphocytes or ≥50% increase in liver and/or spleen size or transformation to a more aggressive histology
Time Frame: At week 9, and post 18 weeks of treatment, then every 3 months for a year and up every 6 months for up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab and Rituximab
Number analyzed (Participants) | 30
Participants
  Complete Remission | 18
  Partial Remission | 12
  Stable Disease | 0
  Progressive Disease | 0

5. Post Hoc Outcome: Best Response in Patients Treated With Alemtuzumab and Rituximab Combination Assessed by NCI-WG 1996 Criteria With Measurements of the Lymph Nodes and Spleen Size by CT Scans
Description: Best Response to treatment, in general is defined as:
  Complete Remission= absence of significant lymphadenopathy and no hepatomegaly/splenomegaly.
  Partial Remission=reduction in lymphadenopathy as defined by the following: (a) 50% decrease in lymph node size by 50% either in the sum products of up to six lymph nodes, or in the largest diameter of the enlarged lymph node(s) detected prior to therapy; (b) no increase in any lymph node, and no new enlarged lymph node; in small lymph nodes (<2cm),and a reduction in the noted pretreatment enlargement of the spleen or liver by 50% or more.
  Stable Disease=not meet criteria for complete/partial remission or progressive disease Progressive Disease=appearance of any new lesion, such as enlarged lymph nodes (1.5cm), splenomegaly, hepatomegaly or other organ infiltrates: (a)50%increase + in greatest diameter of any previous site; (b)50% + increase liver or spleen size.
Time Frame: At week 9, and post-18 weeks then every 3 months for a year and up every 6 months for up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab and Rituximab
Number analyzed (Participants) | 30
Participants
  Complete Remission | 7
  Partial Remission | 14
  Stable Disease | 9
  Progressive Disease | 0

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events (including serious adverse event (SAE) due to hospitalizations) and data was collected, from the time of treatment initiation through 18 weeks of treatment. All cause mortality was collected during 18 weeks of treatment and through 5 years of follow up. Additionally, new cancer SAEs were collected through treatment and through 5 years of follow up.
Arm/Group | Alemtuzumab and Rituximab
All-Cause Mortality (participants affected / at risk) | 4/30
Serious Adverse Events (participants affected / at risk) | 11/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab and Rituximab (N=30)
Possible infection with fever (Infections and infestations) | 2 (2)
Chronic myelogenous leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Multiple myeoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urachal adenocarcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Possible acute renal failure (Renal and urinary disorders) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab and Rituximab (N=30)
Allergic rhinitis (including sneezing,nasal stuffiness,postnasal drip) (General disorders) | 1
Ear pressure/pain (Ear and labyrinth disorders) | 1
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 24
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 18
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 29
Lymphopenia (Blood and lymphatic system disorders) | 30
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 19
Hypotension (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Malaise (General disorders) | 2
Fatigue (General disorders) | 12
Fever (General disorders) | 15
Insomnia (General disorders) | 3
Rigors (General disorders) | 4
Chills (General disorders) | 4
Sweating (General disorders) | 13
Weight loss (General disorders) | 9
Shaking (General disorders) | 1
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 24
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8
Perivascular neutrophilic dermatitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 12
Sun burn (Skin and subcutaneous tissue disorders) | 1
Skin peeling (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 2
Hives (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blotchiness (Skin and subcutaneous tissue disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 4
Anorexia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Mucositis/stomatitis (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Dry lips (Gastrointestinal disorders) | 2
Taste alteration(dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Scratchy throat (Gastrointestinal disorders) | 3
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Lung (pneumonia) (Infections and infestations) | 1
Upper airway infection NOS (Infections and infestations) | 1
Adenovirus (Infections and infestations) | 1
NOS (Infections and infestations) | 2
CMV positive (Infections and infestations) | 5
Edema (Blood and lymphatic system disorders) | 1
:Edema:trunk/genital (Blood and lymphatic system disorders) | 1
Alkaline phosphatase (Metabolism and nutrition disorders) | 9
Transaminase (Metabolism and nutrition disorders) | 11
Bicarbinate high (Metabolism and nutrition disorders) | 1
High GFR (Metabolism and nutrition disorders) | 2
ALT, SGPT (serum glutamic pyruvic transaminase)high (Metabolism and nutrition disorders) | 4
AST, SGOT (serum glutamic oxaloacetic transaminase) high (Metabolism and nutrition disorders) | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 14
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3
High LDH (Metabolism and nutrition disorders) | 6
Increased BUN (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 13
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 24
Glucose, serum-low(hypoglycemia) (Metabolism and nutrition disorders) | 4
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1
Magnesium, serum-low(hypomagnesemia) (Metabolism and nutrition disorders) | 3
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-high(hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low(hypokalemia) (Metabolism and nutrition disorders) | 4
Sodium, serum-high(hypernatremia) (Metabolism and nutrition disorders) | 4
Sodium, serum-low(hyponatremia) (Metabolism and nutrition disorders) | 11
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2
Neuropathy:sensory (Nervous system disorders) | 4
Motor - hand tremors (Nervous system disorders) | 1
Dizziness (Psychiatric disorders) | 4
Mood alteration - Anxiety (Psychiatric disorders) | 1
Mood alteration - Depression (Psychiatric disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Muscle aches (Musculoskeletal and connective tissue disorders) | 1
Pain : ear (Ear and labyrinth disorders) | 1
Abdomen pain NOS (Gastrointestinal disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Hematuria (General disorders) | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
GENERAL- Pain (General disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1
Flashing lights (Eye disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Renal incontinence (Renal and urinary disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 1
Flu-like syndrome (General disorders) | 4
Nasal drip (General disorders) | 1
Nasal congestion (General disorders) | 1
vaginal burning (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes